CLINICAL TRIAL: NCT00679055
Title: An Exploratory Double-Blind, Placebo Controlled, Randomized, 12-Week Oral Dose Study to Evaluate the Effects of MK0736 on Atherosclerotic Disease Biomarkers in Lower Extremity Plaque Excised From Patients With Peripheral Arterial Disease
Brief Title: A Study of How MK-0736 Affects Arterial Plaque (0736-006)(TERMINATED)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: FoxHollow Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0736-006; 2007_600
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-0736 (Experimental): Participants will be orally administered 7 mg of MK-0736 once daily for 12 weeks
  Interventions: Drug: Comparator: placebo (unspecified)
- Placebo (Placebo Comparator): Participants will be orally administered placebo once daily for 12 weeks.
  Interventions: Drug: MK-0736

INTERVENTIONS:
Drug: MK-0736 — MK-0736; 7mg once daily, orally at approximately the same time each morning for 12 weeks.
  Arms: Placebo
Drug: Comparator: placebo (unspecified) — Matching Placebo once daily, orally at approximately the same time each morning for 12 weeks.
  Arms: MK-0736

SUMMARY:
A 12-Week Efficacy Study in participants with Peripheral Arterial Disease. the primary hypothesis is that MK-0736 7 mg administered once daily for 12 weeks will result in a decrease in lower extremity atherosclerotic plaque macrophage content when compared to placebo (an approximate decrease of up to 30% is expected).

ELIGIBILITY:
Inclusion Criteria:

* Participants with peripheral arterial disease
* Participants must be 18 to 85 years of age
* Females must be postmenopausal or sterile

Exclusion Criteria:

* Participans with hepatic, HIV, endocrine, connective tissue, psychiatric disorders or uncontrolled hypertension

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-03-31 (Actual); Primary Completion 2008-08-26 (Actual); Study Completion 2008-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0736-006&kw=0736-006&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-0736 | Placebo
Started | 8 | 6
Completed | 6 | 1
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Other | 0 | 3
Not completed — Study Terminated | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0736 | Placebo | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (7.4) | 70.8 (8.6) | 69.0 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cluster of Differentiation 68 (CD68)
Description: CD68 is a heavily glycosylated transmembrane protein resident to macrophage lysosomes, and is the standard immunohistochemical (IHC) marker for macrophages in human tissues. CD68 protein content as a measure of macrophage number is the most often reported marker in clinical studies of plaque instability. Blood samples were taken to determine the level of CD69 present at baseline (predose Day 1) and again after 12 weeks of study drug administration in participants with peripheral arterial disease of the lower extremity who are scheduled for excision of an atherosclerotic plaque.
Time Frame: Baseline and Week 12
Population: Study terminated early. Planned analyses was not performed.
Arm/Group | MK-0736 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Messenger Ribonucleic Acid (mRNA)
Description: mRNA is a biomarker associated with the inflammatory response. Blood samples were taken to determine the level of mRNA present at baseline (predose Day 1) and again after 12 weeks of study drug administration in participants with peripheral arterial disease of the lower extremity who are scheduled for excision of an atherosclerotic plaque.
Time Frame: Baseline and Week 12
Population: Study terminated early. Planned analyses was not performed.
Arm/Group | MK-0736 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Who Were Discontinued From the Study Due to an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the study drug. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an AE. The percentage of participants who were discontinued from the study due to an AE was summarized.
Time Frame: up to 14 weeks
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: Particpants
Arm/Group | MK-0736 | Placebo
Number analyzed (Participants) | 8 | 6
Particpants | 0 | 1

ADVERSE EVENTS:
Time Frame: up to 14 weeks
Description: All enrolled participants who recieved at least one dose of study drug.
Arm/Group | MK-0736 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/6
Other Adverse Events (participants affected / at risk) | 5/8 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0736 (N=8) | Placebo (N=6)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0736 (N=8) | Placebo (N=6)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0)
Hepatic congestion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated due to lack of recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.